CLINICAL TRIAL: NCT04648592
Title: Impact of Salt Intake on Gut Microbiota, Th17 Immune Response and Endothelial Function in Hypertensive Patients
Brief Title: Salt Intake, Microbiota, Immune Response and Endothelial Function in Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Armando Coca Rojo, Principal Investigator, Hospital Clínico Universitario de Valladolid
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: PI 19-1342
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Hypertension
Keywords: Hypertension; Salt intake
MeSH Terms: conditions — Hypertension | interventions — Diet, Sodium-Restricted; Salts

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blind clinical trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Trial participants, care providers and study investigators will be blinded to assigned interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Low salt diet, aiming at a daily sodium intake of 50 mmol plus oral salt supplements (9 grams) to achieve an overall daily sodium intake of 200 mmol.
  Interventions: Dietary Supplement: Low salt diet plus sodium chloride supplements
- Control (Placebo Comparator): Low salt diet, aiming at a daily sodium intake of 50 mmol plus oral placebo supplements to achieve an overall daily sodium intake of 50 mmol.
  Interventions: Dietary Supplement: Low salt diet plus placebo

INTERVENTIONS:
Dietary Supplement: Low salt diet plus sodium chloride supplements — Patients will receive a low salt diet plus salt supplements.
  Other Names: Salt
  Arms: Intervention
Dietary Supplement: Low salt diet plus placebo — Patients will receive a low salt diet plus placebo.
  Other Names: Placebo
  Arms: Control

SUMMARY:
Hypertension is a significant cardiovascular risk factor which affects 45% of the adult population. Salt intake is essential in the development and progression of hypertension. A reduction in salt intake is associated with a reduction in blood pressure and a 25% lower risk of suffering a cardiovascular event. The mechanisms involved in the association between salt intake and blood pressure are a topic of discussion. Increased salt intake can modify cardiovascular function, inducing endothelial dysfunction, modyfing the activity of the immune system and increasing inflammation or oxidative stress.

In recent years, dietary salt intake has been linked to intestinal depletion of certain genera of bacteria such as Lactobacillus. Tryptophan metabolites formed by these bacteria have been shown to modulate the activity of pro-inflammatory cells such as Th17/CD4+, interleukin 17a producing cells. Studies in animal models have demonstrated that interleukin 17a is able to raise blood pressure by hindering endothelium-dependent vasodilation mechanisms. It is also able to cause sodium and water retention, increase albuminuria, induce renal microvascular injury and vasoconstriction and promote vascular stiffening, cardiac hypertrophy and fibrosis.

The main objective of this trial is to describe the relationship between salt intake, gut commensal microbiota, Th17 activity, endothelial dysfunction and blood pressure evolution in a sample of patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of primary hypertension on treatment for at least 12 months with an ACEI or ARB-II in monotherapy.
* Able to understand the study objectives and to provide written informed consent.

Exclusion Criteria:

* Severe hypertension, defined as a sitting systolic blood pressure ≥200 mmHg, a sitting diastolic blood pressure ≥115 mmHg or a maximum-minimum difference of ≥20 mmHg in systolic blood pressure or ≥10 mmHg in diastolic blood pressure between the right and left arms after three measurements on each arm.
* Suggestive symptoms of secondary hypertension, such as abrupt onset hypertension, age <30 years, advanced end organ damage, new-onset diastolic hypertension in the elderly,
* Treated with antihypertensive drugs other than ACEIs or ARBs.
* Use of drugs that affect diuresis or natriuresis.
* Poorly controlled type 1 or 2 diabetes, defined as a fasting blood glucose ≥200 mg/dl or HbA1c ≥9%.
* History of cardiovascular disease, defined as acute myocardial infarction, ischemic transient attack or stroke, congestive heart failure, peripheral vascular disease or cardiac arrhythmias.
* Chronic obstructive pulmonary disease.
* Liver or kidney disease.
* Pregnant or lactating women.
* Legal incapacity or impossibility to understand the study objectives.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Absolute change in lymphocyte subset counts | 30 days
  Lymphocyte subset counts

SECONDARY OUTCOMES:
Relative change in gut microbiota composition daily total salt | 30 days
  Taxonomic metagenomic analysis, analyzing the composition at the level of family, genus and species. Percentage of variation of each species in each control.
Relative change in body composition assessed by electrical bioimpedance | 30 days
  Percentage of change in total body water, total intracellular water, total extracellular water, fat mass, percentage of fat, lean mass, and muscle-skeletal mass.
Absolute change in peak and average 24h ambulatory blood pressure measurement | 30 days
  24h ambulatory blood pressure measurement
Absolute change in endothelial function | 30 days
  Pulse wave velocity analysis

CONTACTS AND LOCATIONS:
Overall Officials: Armando Coca, MD, MSc, phD, Principal Investigator — Hospital Clínico Universitario Valladolid
Locations (1):
- Hospital Clínico Universitario, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No
Study data will be shared upon reasonable request.